CLINICAL TRIAL: NCT02677272
Title: Factors Predisposing to Inappropriate Transfers of Nursing Home Residents to Emergency Departments
Acronym: FINE
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Agence Régionale de la Santé - Midi Pyrénées (Other Government); Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: RC31/15/7464; 2015-A00723-46 (Other: ID-RCB)
Record Dates: First submitted 2016-01-08; First posted 2016-02-09 (Estimated); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Frail Elderly
Keywords: Nursing home; emergency department; inappropriate transfer; elderly
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Appropriateness of NH resident's transfer to ED

SUMMARY:
According to the data of our nursing homes (NH) research network (REHPA - Gérontopôle Toulouse, 345 nursing home in France), 13.5% of NH residents are hospitalized every 3 months or about 50% per year. These hospitalizations concern for half, transfers to emergency department (ED). Data from the literature and the PLEIAD study, conducted with 300 NH in France, confirm that intense flows between NH and ED. These studies also support the idea that these transfers to ED potentially expose some NH residents to iatrogenic complications, a risk of functional decline, an increased risk of mortality, and generate additional health costs. To transfer to ED residents who will benefit from emergency care and not to transfer to ED residents for whom this transfer generates a higher risk than the expected benefit is the goal to reach to guarantee the better quality of care for NH residents.

Inappropriate transfer to ED may be defined by the absence of somatic emergency and / or palliative care known before transferring to ED and / or the presence of advance directives of non-hospitalization in the resident's file. This is a clinical situation that could be managed by other means that the transfer to ED without loss of opportunity for the patient.

The primary objective of our study is to determine the factors predisposing NH residents to inappropriate transfer to ED.

Our hypothesis is that inappropriate transfers to the ED of NH residents are conditioned by factors accessible to interventions such as the organization of the NH care system or by improving the management of some diseases in NH. Investigators also hypothesize that the cost of inappropriate transfers to the ED is considerable. Acknowledgement of costs generated by inappropriate transfers to ED would allow policy makers to make strategic decisions to improve care system.

DETAILED DESCRIPTION:
This is a retroprospective study conducted in sixteen hospitals in south-west of France. Inclusion will last one year, including 4 periods (one per season) of 7 days (24h / 24, including necessarily each day of the week). All the NH residents admitted in ED will be included. For each resident included, medical and non-medical data will be collected in 4 times: retrospectively before transfer to ED (=T0); and prospectively : at ED (= T1), in hospital services in case the patient is hospitalized (=T2) and at the patient's return to NH (=T3).

At T0 data collected will concern the NH and resident basis medical state, resident's medical state the week before transfer and resident medical state before transfer to ED.

At T3 data collected will concern the resident's return modality and his/her autonomy 7 days after his/her return

Time frame:

between T1 and T3 : mean expected duration will variate from few hours if the resident isn't hospitalized (ED visit) to an average 12.4 days, which is the average length of hospital stay of NH resident hospitalized after a transfer to ED (cf Pleiad study, Rolland 2012) plus 7 days as Investigators will collect T3's data 7 days after the NH resident's return to NH

ELIGIBILITY:
Inclusion Criteria:

* to live in a Nursing Home
* to be directly transferred from the NH to ED
* to have not previously been included in FINE study

Exclusion Criteria:

* to live in structures other than Nursing Home (i.e. sheltered housing, seniors' residences, housing homes, retirement homes, long-term care units)
* to live in the community
* to be transferred to ED from elsewhere than the NH
* to have previously been included in FINE study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients living in Nursing Home admitted in Emergency Department of the hospitals participating in the study during the inclusion period will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1040 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Inappropriate transfer to ED of NH residents | Baseline (T1 = inclusion at ED): retro-prospectively by the group of experts
  Inappropriateness of the NH residents' transfers to ED : the inappropriateness of ED transfers will be determined by the opinion of a group of experts composed of geriatricians, emergency physicians, general practitioners and pharmacists. Inappropriate transfer to ED is defined by the absence of somatic emergency and / or palliative care known before decision to transfer and / or the presence of advance directives of non-hospitalization in the resident's file. This is a clinical situation that could be managed by other means that the transition to ED without loss of opportunity for the resident. To judge the inappropriateness of the transfer to ED, the group of experts will use a rating scale of usual emergencies. Individual and independent rating divergences will lead to a concerted evaluation of the clinical situation by the group.
  Analyse retro-prospectively by the group of experts.

SECONDARY OUTCOMES:
Cost of the NH resident transfer to ED | 6 months before to 6 months after the transfer
  The cost of ED transfers (i.e. appropriate and inappropriate transfers) and the direct medical costs of residents 6 months before and 6 months after the first transfer will be calculated.This work will be lead in partnership with the Regional Direction of the Medical Service of the region and the medico-economic cell of the Medical Information Department of Toulouse University Hospital
Avoidability of the NH resident transfer to ED | Baseline (T1 = inclusion at ED)
  Potentially avoidable transfers to ED: When a transfer is considered appropriate it also can be considered as potentially avoidable if adequate preventive measures were implemented. The Ambulatory Care Sensitive Diagnosis usually used in the literature will be used to characterize the transfers as potentially avoidable. When a transfer is considered inappropriate it is always considered as potentially avoidable. Analyse retro-prospectively by the group of experts.
NH resident's autonomy using Katz'ADL | Change at different time points: T0, T2 (up to 12 days,if concerned) and T3 (7 days after return to NH)
  - Residents' autonomy will be assessed using Katz'ADL at the NH before transfer (T0); at the end of the hospitalization if the resident is concerned (T2), and at the resident's return to ED (T3)
Analysis of Medical prescription, with a focus on psychotropic drug | Change at different time points: T1 (baseline), T2 (up to 12 days,if concerned) and T3 (7 days after return to NH)
  - Medical prescriptions will be collected at inclusion (T1), at the end of the hospitalization if the resident is concerned (T2), and at the resident's return to ED (T3)

CONTACTS AND LOCATIONS:
Overall Officials: Yves ROLLAND, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (16):
- France (16):
  - CH d'Albi, Albi
  - CH d'Auch, Auch
  - CH de Cahors, Cahors
  - CHI Castres Mazamet, Castres
  - CH Ariège Couserans, Foix
  - CH de Gourdon, Gourdon
  - CH Lannemezan, Lannemezan
  - CH Lavaur, Lavaur
  - CH de Lourdes, Lourdes
  - CH Castelsarrasin Moissac, Moissac
  - CH Montauban, Montauban
  - CH Rodez, Rodez
  - CH Saint Gaudens, Saint-Gaudens
  - CHI Val d'Ariège, Saint-Girons
  - Toulouse University Hospital (CHU de Toulouse), Toulouse
  - CH de Bigorre, Vic-en-Bigorre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perrin A, Tavassoli N, Mathieu C, Hermabessiere S, Houles M, McCambridge C, Magre E, Fernandez S, Caquelard A, Charpentier S, Lauque D, Azema O, Bismuth S, Chicoulaa B, Oustric S, Costa N, Molinier L, Vellas B, Berard E, Rolland Y. Factors predisposing nursing home resident to inappropriate transfer to emergency department. The FINE study protocol. Contemp Clin Trials Commun. 2017 Jul 21;7:217-223. doi: 10.1016/j.conctc.2017.07.005. eCollection 2017 Sep. PMID 29696189
- [Result] Rolland Y, Mathieu C, Tavassoli N, Berard E, Laffon de Mazieres C, Hermabessiere S, Houles M, Perrin A, Krams T, Qassemi S, Cambon A, Magre E, Cantet C, Charpentier S, Lauque D, Azema O, Chicoulaa B, Oustric S, McCambridge C, Gombault-Datzenko E, Molinier L, Costa N, De Souto Barreto P. Factors Associated with Potentially Inappropriate Transfer to the Emergency Department among Nursing Home Residents. J Am Med Dir Assoc. 2021 Dec;22(12):2579-2586.e7. doi: 10.1016/j.jamda.2021.04.002. Epub 2021 May 5. PMID 33964225
- [Result] Bouzid W, Cantet C, Berard E, Mathieu C, Hermabessiere S, Houles M, Krams T, Qassemi S, Cambon A, McCambridge C, Tavassoli N, Rolland Y. Exploring Predictive Factors for Potentially Avoidable Emergency Department Transfers: Findings From the FINE Study. J Am Med Dir Assoc. 2024 Apr;25(4):572-579.e1. doi: 10.1016/j.jamda.2023.11.017. Epub 2023 Dec 27. PMID 38159914
- [Result] Dubucs X, Balen F, Charpentier S, Lauque D, De Souto Barreto P, Tavassoli N, Houze-Cerfon CH, Rolland Y. Factors associated with Emergency Medical Dispatcher request and residents' inappropriate transfers from Nursing Homes to Emergency Department. Eur Geriatr Med. 2022 Apr;13(2):351-357. doi: 10.1007/s41999-021-00574-5. Epub 2021 Oct 15. PMID 34652784
- [Derived] Gombault-Datzenko E, Costa N, Mounie M, Tavassoli N, Mathieu C, Roussel H, Lagarrigue JM, Berard E, Rolland Y, Molinier L. Cost of care pathways before and after appropriate and inappropriate transfers to the emergency department among nursing home residents: results from the FINE study. BMC Geriatr. 2024 Apr 19;24(1):353. doi: 10.1186/s12877-024-04946-x. PMID 38641801